CLINICAL TRIAL: NCT04533568
Title: A Randomized-controlled Study; Comparison of the Effectiveness of Intravenous Ibuprofen and Intravenous Dexketoprofen in the Treatment of Migraine-related Headache in the Emergency Department
Brief Title: Ibuprofen in Migraine Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Şeref Kerem Çorbacıoğlu, Associated Professor, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66175679
Record Dates: First submitted 2020-08-22; First posted 2020-08-31 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Migraine Without Aura
Keywords: migraine without migraine; intravenous ibuprofen; intravenous dexketoprofen
MeSH Terms: conditions — Migraine without Aura | interventions — Ibuprofen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ibuprofen (Experimental): 400mg intravenous ibuprofen with 10mg intravenous metoclopramide Hcl in 100ml 0.9% NaCl for 30 minutes.
  Interventions: Drug: Ibuprofen 400 mg
- dexketoprofen (Experimental): 50 mg intravenous dexketoprofen with 10mg intravenous metoclopramide Hcl in 100ml 0.9% NaCl for 30 minutes.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Ibuprofen 400 mg — 400mg intravenous ibuprofen with 10mg intravenous metoclopramide Hcl in 100ml 0.9% NaCl for 30 minutes.
  Arms: ibuprofen
Drug: Dexketoprofen — 50 mg intravenous dexketoprofen with 10mg intravenous metoclopramide Hcl in 100ml 0.9% NaCl for 30 minutes.
  Arms: dexketoprofen

SUMMARY:
In this study, the investigators planned to compare the effectiveness of an intravenous ibuprofen against an intravenous dexketoprofen among patients (18-65 years) who were admitted to the emergency department (ED) with acute migraine-related headaches and diagnosed migraine without aura.

In this study, patients who presented with migraine-related headache to emergency departments will be included in this study. Two different therapy option are created; first, 400mg intravenous ibuprofen with 10mg intravenous metoclopramide Hcl , second, 50 mg intravenous dexketoprofen with 10mg intravenous metoclopramide Hcl.

Patients's headache scores will be measured with visual analog score (VAS) at the pretreatment and post-treatment periods (0. minutes, 30. minutes, and 60. minutes.) 60 minutes after treatment, as a rescue therapy, 100mg tramadol will be given to patients whose headache score does not decrease by more than 50% from pretreatment-VAS score.

ELIGIBILITY:
Inclusion Criteria:

* All the patients aged 18-65 years who had been admitted to the ED for headaches and diagnosed acute migraine-related headache according to the International Classification of Headache Disorders-2018 edition
* Patients whose pre-treatment VAS scores are more than 40 point.
* Patients who give written and verbal consent to include study.

Exclusion Criteria:

* Patients had taken any analgesic drugs or drugs for migraine prophylaxis in the last 6 hours
* Patients had a history of allergy to any of the drugs used in this study
* Patients used any anticoagulant-agents,
* Patients had bleeding diathesis
* patients were pregnant,
* patients were breastfeeding mothers
* Patients who had chronic heart disease, chronic liver disease, and chronic kidney disease
* Patients had peptic ulcer
* Patients had a history of acute akathisia or acute dystonia to metoclopramide hcl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Resolving of Headache at 60 minute | 60 minutes after treatment - Change from Baseline Visual Analog Scale at 60th minutes
  Patients's headache scores will be measured by using Visual Analog Scale (VAS). This scale ranged from 0mm (no pain) to 100mm (worst pain). Measurements will be performed at pre-treatment period and 60th minute after treatments.

SECONDARY OUTCOMES:
Resolving of Headache at 30 minute | 30 minutes after treatment-Change from Baseline Visual Analog Scale at 30th minutes
  Patients's headache scores will be measured by using Visual Analog Scale (VAS). This scale ranged from 0mm (no pain) to 100mm (worst pain). Measurements will be performed at pre-treatment period and 30th minutes after treatments.
Needing of rescue treatment | 60 minutes after treatment
  60 minutes after treatment, as a rescue therapy, 100mg tramadol will be given to patients whose headache pain score - which measured by using Visual Analog Scale (VAS) - does not decrease by more than 50% from pretreatment-VAS score. This scale ranged from 0mm (no pain) to 100mm (worst pain).
Side and adverse effects | From start of performing drug to in the first 24 hours after drug administration
  any side/adverse effects related to study drugs such as hypotension, bradycardia, or anaphylaxis or local adverse effects such as pain or hematoma in the injection area

CONTACTS AND LOCATIONS:
Locations (1):
- Kecioren Training and Research Hospital, Ankara, Turkey (Türkiye)